CLINICAL TRIAL: NCT06546111
Title: Clinical Study to Evaluate the Possible Efficacy and Safety of Diosmin and Hesperidin Combined Therapy in Patients With Helicobacter Pylori Infection
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sadat City University (Other)
Responsible Party: Principal Investigator, Aya Mosaad Zaki Swidan, Demonstrator, Sadat City University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00612/2024
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Diosmin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (placebo group) (Placebo Comparator): Patients will receive standard triple therapy (Omeprazole 20 mg cap PO BID + Clarithromycin 500 mg tab PO BID + Amoxicillin 1000 mg PO BID) and placebo tab PO BID for 14 days
  Interventions: Drug: Placebo
- Group 2 (intervention group) (Experimental): Patients will receive standard triple therapy (Omeprazole 20 mg cap PO BID + Clarithromycin 500 mg tab PO BID + Amoxicillin 1000 mg PO BID) and Diosmin/Hesperidin (Daflon®) 500mg tab PO BID for 14 days.
  Interventions: Drug: Daflon

INTERVENTIONS:
Drug: Placebo — Drug :placebo tab PO BID for 14 days.
  Arms: Group 1 (placebo group)
Drug: Daflon — Daflon 500 mg tab PO BID for 14 days.
  Arms: Group 2 (intervention group)

SUMMARY:
This study intends to assess the possible effectiveness and safety of Diosmin and Hesperidin combination in patients with Helicobacter pylori Infection through evaluating its effect on stool antigen test and serum levels of inflammatory biomarkers as(TNF-A and MDA).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed H. pylori infection through stool antigen test.

  * Patients did not receive prior eradication therapy.
  * Male and female.
  * Age of 18-75 years old.
  * Good mental well-being to clearly understand the study's objectives, advantages and procedures.

Exclusion Criteria:

* Age less than 18 years.

  * Patients with previous H. pylori eradication therapy.
  * Patients with hypersensitivity/allergy to the study medications.
  * Patients with history of using proton pump inhibitor, H2-blocker, antibiotics that affect H.

pylori in the last month.

* Patients with history of using diosmin and/or hesperidin in the last month.
* Patients with history of gastric tumor or gastrointestinal (GI) surgery.
* Patients with concomitant severe disorders; cardiovascular, pulmonary, renal or hepatic, or active malignancy.
* Pregnancy or breastfeeding.
* History of drug misuse or recent alcohol consumption.
* Patients with gall bladder disorders.
* Patients on blood thinning agents (warfarin, clopidogril, aspirin, etc), anticonvulsants (carbamazepine and phenytoin), muscle relaxants (chlorzoxazone) and NSAID (diclofenac) in order to avoid potential pharmacodynamic and pharmacokinetic drug interactions with diosmin.
* Patients on anti-inflammatory drugs and antioxidant drugs.
* Patients with inflammatory conditions (ulcerative colitis, rheumatoid arthritis, etc.).
* Patients with conditions associated with oxidative stress (smoking, COPD, etc.).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Eradication rate of helicobacter pylori infection | At baseline and after 6 weeks of initiation of therapy
  The primary outcome is the improvement of eradication rate of H. pylori infection which is measured by stool antigen test (Negative result).

SECONDARY OUTCOMES:
Inflammatory biomarkers suppression | At baseline and after 6 weeks of initiation of therapy
  The secondary outcome is the change in the measured specific biomarkers (TNF-α which is measured by pg /mL unit), (MDA which is measured by µmol/L)

CONTACTS AND LOCATIONS:
Locations (1):
- National Liver Institute, Shibīn al Kawm, Egypt

IPD SHARING:
Plan to Share IPD: No
Data will be supplied upon a reasonable request